CLINICAL TRIAL: NCT01275235
Title: Metabolic Traits of Adult Sib-pairs Discordant for Intrauterine Diabetes Exposure.
Brief Title: Exposure to Type II Diabetes for Two Siblings With the Same Parents
Acronym: T2DM
Status: Terminated | Type: Observational
Why Stopped: We were unable to recruit enough sibling pairs in a timely manner.
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Darcy Johannsen, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 10016
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Whole blood, urine and muscle cell.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Exposure to Type II Diabetes for two siblings: Two sibling pairs with the same parents, between the ages of 20 to 34 in the Baton Rouge Area, having mother with diabetes while pregnant with one.

SUMMARY:
Individuals with a family history of type 2 diabetes mellitus (T2DM) are known to be at greater risk for the disease, and studies have shown that how the body responds to insulin, how the muscle creates energy, and the amount of fat stored inside skeletal muscle are often different in these individuals at a young age compared to people without a family history of the disease. The tendency to develop T2DM is influenced strongly by genetics; however, exposure to the surrounding environment may also play a role. The exposure to a diabetic environment while in the womb represents an altered nutritional exposure (high levels of circulating sugar, or glucose) that may affect how tissues important in regulating energy metabolism, such as the pancreas, liver, and skeletal muscle, develop. the purpose of this study is to measure sensitivity to insulin, energy expenditure, fat content of the abdomen and skeletal muscle function in young adult sibling pairs who were raised together but who are discordant for intrauterine exposure to diabetes (i.e., the mother did ot have diabetes during pregnancy with the older sibling, but did have diabetes during pregnancy with the younger sibling).

DETAILED DESCRIPTION:
A one-time testing comprising of 2 days (32 consecutive hours). A medical history and physical including questions about medications, health status and symptoms are acquired at the fasting screening visit. Both siblings must meet all study eligibility requirements to be enrolled into the study. If enrolled for the 2 days, you will be in a metabolic chamber, dual energy x-ray absorptiometry (DXA) scan, biopsy, oral glucose tolerance test, and magnetic resonance imaging (MRI).

* Metabolic chamber is a room is a sophisticated system that allows your oxygen / carbon dioxide exchange to be measured, thereby showing the number of calories you are burning.
* DXA is a scan that measure the amount of bone, muscle, and fat in your body.
* Biopsy is a procedure to sample muscle cells from underneath the skin.
* OGTT is Oral Glucose Tolerance Test from an IV line for blood samples once you drink a sugar solution consisting of glucose.
* MRI scan is to measure the amount of fat in your abdomen around the organs and underneath the skin.

ELIGIBILITY:
Inclusion Criteria:

* You are one of a sibling pair with the same mother and father, and your mother had diabetes (gestational or type 2) while she was pregnant with the younger sibling but not the older sibling.
* Your sibling is willing to participate in the study.
* You are between the ages of 20 and 34 years (inclusive)
* Your body mass index is between 20 and 29 Kg/m2 inclusive (this is a number calculated for your height and weight and indicates that you are either normal weight or overweight, but not obese).
* You are healthy as assessed by medical history and standard physical examination
* You are weight stable (your body weight has not changed .6.5 lbs over the last 3 months).
* You do not smoke
* You provide written informed consent to participate in the study.
* You are willing to stay overnight one time at the Pennington Center.
* You have low physical activity (< 100 min of exercise per week).

Exclusion Criteria:

* You were born prematurely (<37 weeks of pregnancy)
* You are currently taking medication that may influence your body weight or metabolism.
* You have heart disease, lung disease, liver disease, blood disease, kidney disease, type 1 or 2 diabetes, or any other disease that in the opinion of the doctor might make you ineligible.

Ages: 20 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Risk of type 2 diabetes mellitus (T2DM) | 2 days
  The purpose is to measure sensitivity to insulin, energy expenditure, fat content of the abdomen and skeletal muscle function in young adult sibling pairs who were raised together but who are discordant for intrauterine exposure to diabetes (i.e., the mother did not have diabetes during pregnancy with the older sibling, but did have diabetes during pregnancy with the younger sibling).

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Johannsen, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Background] Warram JH, Martin BC, Krolewski AS, Soeldner JS, Kahn CR. Slow glucose removal rate and hyperinsulinemia precede the development of type II diabetes in the offspring of diabetic parents. Ann Intern Med. 1990 Dec 15;113(12):909-15. doi: 10.7326/0003-4819-113-12-909. PMID 2240915
- [Derived] Lam YY, Redman LM, Smith SR, Bray GA, Greenway FL, Johannsen D, Ravussin E. Determinants of sedentary 24-h energy expenditure: equations for energy prescription and adjustment in a respiratory chamber. Am J Clin Nutr. 2014 Apr;99(4):834-42. doi: 10.3945/ajcn.113.079566. Epub 2014 Feb 5. PMID 24500151